CLINICAL TRIAL: NCT04080323
Title: Effect of a Single Preoperative Dose of Vaginal Dinoprostone on Intraoperative Blood Loss During Abdominal Hysterectomy:a Randomized Controlled Trial
Brief Title: Single-dose Vaginal Dinoprostone and Hysterectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: dinoprostone hysterectomy
Record Dates: First submitted 2019-09-04; First posted 2019-09-06 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Hysterectomy
MeSH Terms: interventions — Dinoprostone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dinoprostone 3 mg (Experimental): 60 minutes before the surgery 3 mg of dinoprostone inserted vaginally
  Interventions: Drug: Dinoprostone 3 mg
- placebo (Placebo Comparator): 60 minutes before the surgery 1 tablet of placebo inserted vaginally
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Dinoprostone 3 mg — 1 vaginal tablet of 3mg dinoprostone 60 minutes before surgery
  Arms: dinoprostone 3 mg
Drug: placebo — 1 vaginal tablet of placebo 60 minutes before surgery
  Arms: placebo

SUMMARY:
In this study, we will assess the efficacy of dinoprostone in minimizing blood loss during hysterectomy when used as a single preoperative dose via the vaginal route. The reduction of blood flow may be due to the combined effect of myometrial contraction and vasoconstrictive effect

ELIGIBILITY:
Inclusion Criteria:

* • Patients presenting for hysterectomy for any benign indication including uterine fibroids.

  * Age ≥ 18 years
  * Pre-operative hemoglobin >8 g/dl
  * Willing to have dinoprostone or a placebo prior to hysterectomy
  * Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* • Patients with known or suspected endometrial/ovarian/cervical cancer.

  * Patients undergoing hysterectomy for endometrial hyperplasia or cervical dysplasia.
  * Patients currently undergoing treatment for any type of cancer.
  * Patients with known bleeding/clotting disorders or a history of thromboembolism (including deep venous thrombosis or pulmonary embolism)
  * History of allergic reactions to dinoprostone.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 118 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
decrease blood loss during hysterectomy | intraoperative
  decrease blood loss during hysterectomy in ml

SECONDARY OUTCOMES:
postoperative hemoglobin level | 24 hours
  postoperative hemoglobin level in gm/dl

CONTACTS AND LOCATIONS:
Overall Officials: AHMED SAMY, Study Director — Cairo University; ayman taher, MD, Principal Investigator — Cairo University; ahmed S Ali, Principal Investigator — faculty of medicine al-azhar university
Locations (1):
- Ahmed Samy, Giza, Egypt